CLINICAL TRIAL: NCT02685566
Title: A Multi-Reader Multi-Case Controlled Clinical Trial to Assess the Adequacy of the Fujifilm Full Field Digital Mammography (FFDM) and Digital Breast Tomosynthesis (DBT) Reader Training Program - A Pilot Study
Brief Title: Multi-Reader Multi-Case Controlled Clinical Trial to Assess the Fujifilm FFDM and DBT Reader Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FMSU2013-004F
Record Dates: First submitted 2015-08-17; First posted 2016-02-18 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FFDM Plus DBT (Experimental): Breast Images with FFDM and DBT
  Interventions: Device: FFDM Plus DBT
- Full-Field Digital Mammography (Active Comparator): Breast Images with FFDM alone
  Interventions: Device: FFDM

INTERVENTIONS:
Device: FFDM Plus DBT — FujiFilm Aspire Cristalle System
  Arms: FFDM Plus DBT
Device: FFDM — FujiFilm Aspire Cristalle System
  Arms: Full-Field Digital Mammography

SUMMARY:
The purpose of this pilot is to assess the adequacy of the Fujifilm DBT Reader Study Training program to ensure that Readers participating in the Fujifilm DBT pivotal trial are properly trained in the reading and interpretation of FFDM and DBT images.

DETAILED DESCRIPTION:
For this reader study, radiologists review images obtained via protocol FMSU2013-004A. They review both FFDM alone and FFDM + DBT images, and provide a BI-RADS and POM for each. The radiologists performance metrics for the following modalities will be evaluated: FFDM and FFDM + DBT.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects participating in FMSU004A protocol with known clinical status

Exclusion Criteria:

* Subjects with unknown clinical status not participating in FMSU004A protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Uzenoff, Study Director — Fujifilm Medical Systems USA, Inc.
Locations (5):
- United States (5):
  - Scottsdale Medical Imaging, Limited (SMIL), Scottsdale, Arizona
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Elizabeth Wende Breast Care, LLC (EWBC), Rochester, New York
  - University of North Carolina - at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 100 breast screening and diagnostic cases selected for this study, were obtained from the FMSU2013-004A acquisition study. The statistician randomly selected cases to provide a distribution of density, finding types, etc.
Pre-assignment Details: Each radiologist read all 100 cases as FFDM only and FFDM+DBT(100 cases multiplied by 2 modalities = 200 reads) with a 4 week washout period between the 2 sessions.
Groups:
- FFDM Plus DBT, Then FFDM Only: Readers to read half of the FFDM plus DBT images followed by half of the FFDM only images at each of the 2 sessions. There was a 4 week memory washout period between the 2 sessions.
- FFDM Only, Then FFDM Plus DBT: Readers to read half of the FFDM only images followed by half of the FFDM plus DBT images at each of the 2 sessions. There was a 4 week memory washout period between the 2 sessions.
Period: First Reading Session
Arm/Group | FFDM Plus DBT, Then FFDM Only | FFDM Only, Then FFDM Plus DBT
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: 4 Week Memory Washout Period
Arm/Group | FFDM Plus DBT, Then FFDM Only | FFDM Only, Then FFDM Plus DBT
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Second Reading Session
Arm/Group | FFDM Plus DBT, Then FFDM Only | FFDM Only, Then FFDM Plus DBT
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 100 study participants (resulting in 200 images) in total who had their images reviewed by 6 radiologist readers. Images were acquired under acquisition study FMSU2013-004A.
Groups:
- All 100 Cases/Study Participants: Each case contributed 2 sets of images: FFDM only as well as DBT plus FFDM. Therefore there were 200 reads acquired from the 100 cases/participants.
Arm/Group | All 100 Cases/Study Participants
Number analyzed (Participants) | 100
Age, Continuous [Median (Standard Deviation); unit: years] | 58 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 87
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Assessing Adequacy of Training - Cancer Detection Threshold & Recall Rate
Description: This endpoint was evaluated qualitatively. Reported the number of readers meeting the Pass Criteria on the final FFDM plus DBT assessment case set, which requires adequate performance in cancer cases (detection rate) as well as non-cancer cases (recall rate). Per-subject BI-RADS, POM and recall scores were derived. Credit was only given for identifying a subject with cancer if the reader marked findings in at least one location with cancer. Findings that did not match the location of a malignant lesion were ignored for cancer cases in the per-subject analyses.
Time Frame: 4 weeks
Population: The study employed a fully factorial, counterbalanced crossover design in which all readers reviewed images from all cases in two visits separated by a memory washout period of approximately 4 weeks. Each reader read half FFDM cases and half FFDM + DBT cases during each of 2 visits.
Measure: Mean (95% Confidence Interval); unit: probability
Groups:
- FFDM Plus DBT: Breast Images with FFDM and DBT FFDM Plus DBT: FujiFilm Aspire Cristalle System.
  This endpoint will be evaluated qualitatively. The Pass Criteria require adequate performance in non-cancer cases (recall rate) and in cancer cases (detection rate).
- Full-Field Digital Mammography (FFDM): Breast Images with FFDM alone FFDM: FujiFilm Aspire Cristalle System.
  This endpoint will be evaluated qualitatively. The Pass Criteria require adequate performance in non-cancer cases (recall rate) and in cancer cases (detection rate).
Arm/Group | FFDM Plus DBT | Full-Field Digital Mammography (FFDM)
Number analyzed (Participants) | 100 | 100
probability | .805 [0.701 to 0.910] | 0.756 [0.646 to 0.867]

2. Secondary Outcome: Area Under Curve (AUC) ROC (Receiver Operating Characteristic) Based on Per-subject Probability of Malignancy (POM) Scores Requiring Correct Lesion Localization.
Description: The magnitude and direction of differences between performance metrics for the two modalities, and variance components and correlations that would influence sample size and case mix for the pivotal reader study (FMSU2013-004G) comparing performance metrics between the two modalities, obtained using established methods for analysis of MRMC (multi-reader, multi-case) studies. The statistician estimated AUC's for each reader in each review condition based on per-subject POM scores requiring correct lesion localization. Statistician performed MRMC comparison of AUC's between reading conditions using the MRMC analysis of variance (ANOVA) method.
Time Frame: 5 weeks
Measure: Mean (95% Confidence Interval); unit: Probability
Groups:
- Full-Field Digital Mammography (FFDM): Breast Images with FFDM alone
  FFDM: FujiFilm Aspire Cristalle System
Arm/Group | FFDM Plus DBT | Full-Field Digital Mammography (FFDM)
Number analyzed (Participants) | 100 | 100
Probability | 0.805 [0.701 to 0.910] | 0.777 [0.659 to 0.894]

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: There were no AE's expected for this study, as it was a radiologist reader study utilizing retrospective imaging. No study subjects were on-site for this retrospective review. No Adverse Events to report.
Arm/Group | FFDM Plus DBT | Full-Field Digital Mammography
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No